CLINICAL TRIAL: NCT01602094
Title: Immunity to Measles Virus in the Thai Population Age 18-30 Years and Predictive Factors
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Queen Saovabha Memorial Institute (Other)
Responsible Party: Principal Investigator, Jaruboot Angsanakul, Jaruboot Angsanakul, Queen Saovabha Memorial Institute
Other Study IDs: TAI5501
Record Dates: First submitted 2012-05-16; First posted 2012-05-18 (Estimated); Last update posted 2012-05-18 (Estimated); Status verified 2012-05

CONDITIONS: Measles
Keywords: measles; antibody; prevalence; predictors; Donor of National Blood Centre, The Thai Red Cross Society who age 18-30 years old; Measles antibody levels; Predictors of adequate measles antibody levels and inadequate measles antibody levels
MeSH Terms: conditions — Measles

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Each participant will be taken blood sample approximately 8 ml. The blood sample will be centrifuged and kept as serum. The serum will be kept under - 20 degree Celsius. Then, all serum will be tested by ELISA.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Adequate antimeales antibody levels: ELISA test OD > 0.1
- Inadequate measles antibody levels: ELISA test OD < 0.1

SUMMARY:
Prevalence of participants who have protective immunity to measles virus is less than ninety percent.

Predictor of adequate measles antibody levels include the following :

* History of measles infection
* History of complete measles primary immunization( 2 doses with at least 1 month interval after age of 9 months)
* History of measles exposure

Predictor of inadequate measles antibody levels include the following :

* Born outside Thailand
* History of staying outside Thailand for long time in childhood
* Living in the rural area for a long period in childhood
* Fail to participate school system on time

ELIGIBILITY:
Inclusion Criteria:

* Age 18-30 years old

Exclusion Criteria:

* Last measles vaccination less than 10 years of age
* Immunocompromised host including congenital immune defect, splenectomy or splenic dysfunction, history of suspect HIV exposure, taking immunosuppressant
* Receiving blood or blood product within 3 months
* Receiving others vaccinations or immunoglobulins or any medication that possibly decrease immune response

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Health Thai participant age 18-30 years old.
Sampling Method: Non-Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2012-07; Primary Completion 2013-01 (Estimated); Study Completion 2013-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jaruboot Angsanakul, M.D., Principal Investigator — Queen Saovabha Memorial Institute
Locations (1):
- Queen Saovabha Memorial Institute, Bangkok, Bangkok, Thailand

REFERENCES:
- See also: Contact information — http://www.saovabha.com/en/contactus.asp